CLINICAL TRIAL: NCT05617378
Title: Exploring the Risk Factors for Colorectal Cancer in Our General Population Using Asian Pacific Screening Score: a Survey From Pakistan
Status: Completed | Type: Observational
Sponsor: Sindh Institute of Urology and Transplantation (Other)
Responsible Party: Principal Investigator, Murk Niaz, Medical Officer, Sindh Institute of Urology and Transplantation
Other Study IDs: CRC Survey
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms
Keywords: colorectal carcinoma; Pakistan
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Pakistan, due to the lack of a National based cancer registry exact number of CRC cases is unknown. However, minimal data that is present in literature shows an increase in CRC cases with a concerning increase in incidence in younger age groups11. This makes it pertinent to understand current pattern of CRC and its risk factors from a local perspective. This will direct future strategies in an attempt to reduce the incidence and mortality associated with CRC in our general population.

ELIGIBILITY:
Inclusion Criteria:

* Individuals visiting SIUT as attendants to the patients visiting outpatient department or admitted in hospital.

Exclusion Criteria:

* Attendants / whose patients visit GI, colon and oncology OPD outpatient department or admitted in GI wards.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: attendants to the patients visiting outpatient department or admitted in hospital.
Sampling Method: Probability Sample
Enrollment: 558 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Risk factor | 1 year
  evaluate internationally validated risk factors for colorectal cancer in our general population using a questionnaire based on the modified Asian Pacific Colorectal Screening score.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Shadab Khan, Principal Investigator — Sindh Institute of Urology and Transplantation; Bushra Shirazi, Study Chair — Sindh Institute of Urology and Transplantation; Muhammad Arsalan Khan, Study Chair — Sindh Institute of Urology and Transplantation
Locations (1):
- Sindh Institute of Urology and Transplantation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No